CLINICAL TRIAL: NCT03704220
Title: Safety and Feasibility of Anti-thrombotic Monotherapy With the HeartMate 3 LVAS: A Single Center Prospective Controlled Study
Brief Title: Anti-thrombotic Monotherapy With the HeartMate 3 LVAS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Institute for Clinical and Experimental Medicine (Other Government)
Collaborators: Abbott (Industry)
Responsible Party: Principal Investigator, Prof. Ivan Netuka, MD, Ph.D., Chairman of the Department of Cardiovascular Surgery, Institute for Clinical and Experimental Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Version1.0
Record Dates: First submitted 2018-10-10; First posted 2018-10-12 (Actual); Last update posted 2020-08-04 (Actual); Status verified 2020-08

CONDITIONS: Heart Failure; Cardiovascular Diseases
Keywords: Single anti-thrombotic therapy; Mechanical circulatory support
MeSH Terms: conditions — Heart Failure; Cardiovascular Diseases | interventions — Warfarin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single anti-thrombotic treatment (Other): Single anti-thrombotic treatment
  Interventions: Drug: Warfarin

INTERVENTIONS:
Drug: Warfarin — Removal of anticoagulation with warfarin

SUMMARY:
The purpose of this study is to obtain a single-center safety and feasibility data on patients managed with a single anti-thrombotic therapy and the incidence of thrombotic adverse events associated with HeartMate 3 LVAS therapy.

DETAILED DESCRIPTION:
Patients implanted with the HeartMate 3 LVAS in whom at least 6 months reduced anticoagulation therapy (INR range 1.5-1.9 along with antiplatelet therapy) has been accomplished safely will be screened for participation in the study. If inclusion criteria are met, patients will be transitioned to a single anti-thrombotic therapy with Acetylsalicylic Acid (ASA) and anticoagulation with warfarin will be removed. ASA will be administered in a minimum dose of 100 mg per day with dosage adjustments based on VerifyNow testing up to a maximum of 200 mg daily. The primary endpoint will be analyzed at 90 days after initiation of the single antiplatelet therapy.

ELIGIBILITY:
Inclusion Criteria:

* patients implanted with HeartMate 3 LVAS irrespective of intended goal of treatment of bridge to transplant or destination therapy
* 6 months or more on reduced anti-coagulation regimen (target INR 1.5-1.9) free of thromboembolic and thrombotic complications
* evidence of forward flow across the aortic valve (with aortic valve opening of at least 1:2 per cardiac cycle) at baseline echocardiography (ECHO) or after the speed optimization without a significant progression of heart failure based on a biomarker and complex clinical assessment follow-up

Exclusion Criteria:

* absence of an informed consent
* presence of any prosthetic valve
* known history of major thrombotic event e.g. DVT
* known history of stroke
* left atrial appendage in patients with atrial fibrillation or flutter not addressed by resection or exclusion at a time of the implant
* evidence of any intracardiac thrombus
* any clinical indication for use of long-term warfarin anticoagulation (e.g. known genetic thrombotic mutation, malignancy)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2018-08-16 (Actual); Primary Completion 2021-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
survival free rate of thromboembolic events | 90 days
  Determination of survival free of thromboembolic events (i.e. pump thrombosis or any ischemic stroke) using only a single antithrombotic therapy with Acetylsalicylic Acid.

SECONDARY OUTCOMES:
Adverse Events | 90 days
  Adverse events rates per INTERMACS definitions.

CONTACTS AND LOCATIONS:
Locations (1):
- Institute for Clinical and Experimental Medicine, Prague, Prague 4, Czechia

REFERENCES:
- [Background] Mehra MR, Goldstein DJ, Uriel N, Cleveland JC Jr, Yuzefpolskaya M, Salerno C, Walsh MN, Milano CA, Patel CB, Ewald GA, Itoh A, Dean D, Krishnamoorthy A, Cotts WG, Tatooles AJ, Jorde UP, Bruckner BA, Estep JD, Jeevanandam V, Sayer G, Horstmanshof D, Long JW, Gulati S, Skipper ER, O'Connell JB, Heatley G, Sood P, Naka Y; MOMENTUM 3 Investigators. Two-Year Outcomes with a Magnetically Levitated Cardiac Pump in Heart Failure. N Engl J Med. 2018 Apr 12;378(15):1386-1395. doi: 10.1056/NEJMoa1800866. Epub 2018 Mar 11. PMID 29526139
- [Background] Netuka I, Ivak P, Tucanova Z, Gregor S, Szarszoi O, Sood P, Crandall D, Rimsans J, Connors JM, Mehra MR. Evaluation of low-intensity anti-coagulation with a fully magnetically levitated centrifugal-flow circulatory pump-the MAGENTUM 1 study. J Heart Lung Transplant. 2018 May;37(5):579-586. doi: 10.1016/j.healun.2018.03.002. Epub 2018 Apr 11. PMID 29655662
- See also: Evaluation of low-intensity anti-coagulation with a fully magnetically levitated centrifugal-flow circulatory pump-the MAGENTUM 1 study — https://doi.org/10.1016/j.healun.2018.03.002